CLINICAL TRIAL: NCT04428944
Title: Strategies for Catheter Ablation of Persistent Atrial Fibrillation: a Randomized, Comparative Study
Brief Title: STrategies for Catheter Ablation of peRsistent Atrial Fibrlllation
Acronym: STARAF3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Atul Verma, Cardiologist electrophysiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-33-2021-2805
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PV antral isolation alone (PVAI) (Active Comparator): PV antral isolation alone (PVAI)
  Interventions: Procedure: Wide Circumferential Pulmonary Vein Antrum Isolation (PVAI)
- PV antral isolation plus ablation of drivers (Active Comparator): PV antral isolation plus ablation of drivers (PVAI+drivers)
  Interventions: Procedure: Pulmonary Vein Antrum Isolation Plus Driver Ablation (PVAI+drivers)
- PV antral isolation plus isolation of posterior wall (Active Comparator): PV antral isolation plus isolation of LA posterior wall (PVAI+Box)
  Interventions: Procedure: Pulmonary Vein Antrum Isolation Plus Box Isolation of Posterior Wall (PVAI+box)

INTERVENTIONS:
Procedure: Wide Circumferential Pulmonary Vein Antrum Isolation (PVAI) — Standard PVI
  Arms: PV antral isolation alone (PVAI)
Procedure: Pulmonary Vein Antrum Isolation Plus Driver Ablation (PVAI+drivers) — Standard PVI + Ablation of drivers in LA and RA
  Arms: PV antral isolation plus ablation of drivers
Procedure: Pulmonary Vein Antrum Isolation Plus Box Isolation of Posterior Wall (PVAI+box) — Standard PVI + Electrical isolation of the posterior wall of the left atrium
  Arms: PV antral isolation plus isolation of posterior wall

SUMMARY:
The objective of this study is to compare the efficacy of three different ablation strategies in patients with persistent AF:

1. PV antral isolation alone (PVAI)
2. PV antral isolation plus ablation of drivers (PVAI+drivers)
3. PV antral isolation plus isolation of posterior wall (PVAI+box) All three strategies will employ contemporary catheter ablation technology using more efficient open irrigated tip cooling and contact force sensing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Patients undergoing first-time ablation procedure for AF
3. Patients with persistent AF defined as a sustained episode more than 3 months but less than three years
4. Patients with symptomatic AF - symptomatic patients are those who have been aware of their AF at any time within the last 5 years prior to enrolment. Symptoms may include, but are not restricted to, palpitations, shortness of breath, chest pain, fatigue, left ventricular dysfunction, or other symptoms or any combination of the above
5. Patients whose AF has been refractory to at least one antiarrhythmic drug
6. At least one episode of AF must have been documented by ECG, holter, loop recorder, telemetry, trans-telephonic monitor or implanted device within the last 2 years from enrolment
7. Patients must be able and willing to provide written informed consent to participate in the study

Exclusion Criteria:

1. Patients with paroxysmal AF (no episodes lasting > 7 days)
2. Patients with early persistent AF, sustained episode ≤ 3 months
3. Patients with very long lasting persistent AF (episodes lasting > 3 years)
4. Patients with CHA2DS2-VASc score of 0.
5. Patients for whom cardioversion or sinus rhythm will never be attempted/pursued
6. Patients with AF felt to be secondary to an obvious reversible cause
7. Patients with contraindication to oral anticoagulation or systemic anticoagulation with heparin
8. Patients with left atrial diameter > 60 mm in the parasternal long axis view
9. Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from documented atrial arrhythmia ≥ 30 seconds at 18 months after one ablation procedure on or off antiarrhythmic medications (AAM). | 18 months

SECONDARY OUTCOMES:
Freedom from documented AF > 30 seconds at 18 months after one procedure on or off AAM | 18 months
Freedom from documented AF > 30 seconds at 18 months after one or more procedures on or off AAM | 18 months
Freedom from documented atrial arrhythmia > 30 seconds at 18 months after one or more procedures on or off AAM | 18 months
Freedom from documented AF > 30 seconds at 18 months after one procedure off AAM | 18 months
Freedom from documented atrial arrhythmia > 30 seconds at 18 months after one procedure off AAM | 18 months
Freedom from documented AF > 30 seconds at 18 months after one or more procedures off AAM | 18 months
Freedom from documented atrial arrhythmia > 30 seconds after one or more procedures off AAM | 18 months
Freedom from documented symptomatic AF > 30 seconds at 18 months after one procedure on or off AAM | 18 months
Freedom from documented symptomatic atrial arrhythmia > 30 seconds after one procedure on or off AAM | 18 months
Each of the above success measures stratified by CHA2DS2-VASc score | 18 months
Incidence of peri-procedural complications including stroke, PV stenosis, cardiac perforation, esophageal injury, phrenic nerve palsy, and death | 18 months
Procedure duration | 18 months
Fluoroscopy time (dose) | 18 months
Radiofrequency time | 18 months
Number of repeat procedures | 18 months
Effect of each strategy on AF cycle length changes and AF termination | 18 months
Correlation of acute AF termination on long-term procedural outcome | 18 months
Quality of life measurements during follow-up using AFEQT questionnaire | 6-12-18 months
  AFEQT questionnaires will be used at baseline, 6, 12 and 18 months
Quality of life measurements during follow-up using SF12 questionnaires | 6-12-18 months
  SF36 questionnaires will be used at baseline, 6, 12 and 18 months
Change in AF burden post-ablation procedure (% of time in AF) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, Dr., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Laurent Macle, Dr., Principal Investigator — Montreal Heart Institute
Locations (32):
- Brigham & Women'S Hosptial Inc., Boston, Massachusetts, United States
- Australia (4):
  - Canberra Heart Rhythm Foundation, Garran, Australian Capital Territory
  - Royal Adelaide Hospital and Cardiovascular Centre, Adelaide
  - Alfred Health, Melbourne
  - Royal Melbourne Hospital, Parkville
- Austria (2):
  - Medical University of Graz, Graz
  - Ordensklinikum Linz GmbH, Linz
- Belgium (3):
  - OLV Hospital Aalst, Aalst
  - Antwerp University Hospital (UZA), Edegem
  - AZ Sint-Jan, Ruddershove
- Canada (11):
  - University of Calgary Foothills, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Colombia
  - St. Paul's Hospital, Vancouver, BC, Vancouver, British Colombia
  - Royal Jubilee Hospital, Victoria, British Colombia
  - Hamilton General Hospital, Hamilton, Ontario
  - Southlake Regional Health Center, Newmarket, Ontario
  - Laurent Macle, Montreal, QC - Québec
  - MUHC, McGill University Health Centre, Montreal, Quebec
  - University of Ottawa Heart Institute, Ottawa, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ), Québec, Quebec
  - Hôpital Fleurimont, CHUS, Sherbrooke, Quebec
- France (3):
  - Hospital St-Joseph, Marseille
  - Institut Mutualiste Montsouris, Paris
  - Clinique du Tonkin, Villeurbanne
- Ospedale Generale Regionale F. Miulli, Acquaviva delle Fonti, Italy
- Japan (6):
  - Dokkyo Medical University Koshigaya Hospital, Koshigaya, Saitama
  - Juntendo University Hospital, Bunkyo City, Tokyo
  - National University Corporation Kobe University, Chūōku
  - Jikei University School of Med, Tokyo
  - Minamino Cardiovascular Hospital, Tokyo
  - Nihon University School of Medicine, Tokyo
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No